CLINICAL TRIAL: NCT06437899
Title: Evaluation of Efficacy and Patient Satisfaction Using Local Anaesthesia Versus Sedoanalgesia for Intradetrusor Botulinum-Toxin A Injection for the Treatment of Idiopathic Overactive Bladder: a Randomized Controlled Non-inferiority Trial
Brief Title: Evaluation of Efficacy and Patient Satisfaction of Local Anaesthesia Versus Sedoanalgesia for Botox (R) Injection in the Urinary Bladder for the Treatment of Idiopathic Overactive Bladder
Acronym: LA vs SA
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital LKH Hochsteiermark - Leoben (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21346; AUB (Other: AUB - Arbeitsgemeinschaft für Urogynäkologie Österreich)
Record Dates: First submitted 2024-03-30; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Overactive Bladder
Keywords: overactive bladder; botulinum toxin A; local anaesthesia
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- local anaesthesia (Active Comparator)
  Interventions: Drug: intravesical botulinum toxin A injection unter local anaesthesia
- sedoanalagesia (Active Comparator)
  Interventions: Drug: intravesical botulinum toxin A injection unter local anaesthesia

INTERVENTIONS:
Drug: intravesical botulinum toxin A injection unter local anaesthesia — Arm1: Botulinum toxin A injection under local anesthesia according to standard protocol:
  Retrograde filling of the empty urinary bladder with a 1:1 mixture of 50 ml lidocaine 1% mixed with 50 ml sodium bicarbonate 8.4%, leave the local anesthetic mixture in the bladder for 15 minutes.
  Transurethral, intravesical injection of a total of 100IE botulinum toxin A dissolved in 10 ml NaCl 0.9% into the detrusor at 10 points using a rigid 70 degree cystoscope
  Arm 2: botulinum toxin A injection in sedoanalgesia according to the anesthesia standard protocol:
  Intravenous administration of remifentanil (0.05-0.15µg/kg/min) and propofol. Transurethral, intravesical injection of a total of 100IE botulinum toxin A dissolved in 10ml NaCl 0.9% into the detrusor.

SUMMARY:
Patients with symptoms of overactive bladder suffer from frequent micturition, urinary incontinence and recurrent urinary tract infections. Intravesical injections with botulinum toxin A can be used as a second-line therapy for this purpose.

Intravesical botulinum toxin A injections can be performed under general anesthesia, regional anesthesia, sedoanalgesia and local anesthesia. Which form of anesthesia is used varies greatly from region to region.

As these patients are often elderly and morbid, the lowest-risk and least stressful anesthesia method should be used. The lowest-risk anesthesia method that can be used is local anesthesia. Currently, there are no guidelines that describe the use of standardized protocols for local anesthesia.

The aim of this study is to show that the use of local anesthesia in this context is not inferior to the use of sedoanalgesia.

All patients with overactive bladder symptoms who fulfill the inclusion criteria and present at the Urogynecology Outpatient Clinic of the Department of Gynecology and Obstetrics at the LKH Hochsteiermark in Leoben within 24 months will be invited to participate in the study.

The main outcome measure is pain, secondary outcome measures are quality of life, patient satisfaction, incontinence score, operation time and length of stay in the recovery room, acceptance of repeating the procedure under local anesthesia, satisfaction with the type of anesthesia method, side effects/complications and duration of inpatient stay.

The study will be randomized into 2 arms (local anesthesia/sedoanalgesia) with a 1:1 ratio to carry out the intravesical injection with botulinum toxin A.

DETAILED DESCRIPTION:
Urinary urgency symptoms with frequent micturition, urinary incontinence, nocturia and recurrent urinary tract infections are typical complaints of women with symptoms of an overactive bladder. The level of suffering is usually very high. Social withdrawal, depressive moods, frequent antibiotic use and financial burdens due to the increased need for incontinence products can be the result. In accordance with the guideline-based treatment of idiopathic overactive bladder, intravesical injection of botulinum toxin A can be offered after unsuccessful conservative first-line and second-line treatment. Intravesical injection of botulinum toxin A has been approved for the treatment of idiopathic overactive bladder in Austria since 2013. Botulinum toxin A is a registered drug in Austria and is used for injection into the detrusor with 100IE according to its approval indication.

Intravesical botulinum toxin A injections can be performed under general anesthesia, regional anesthesia, sedoanalgesia and local anesthesia. Which form of anesthesia is used varies greatly from region to region. The effectiveness of botulinum toxin A is limited in time. Injections are repeated on average after 6-12 months. Patients are often older and often have comorbidities. Due to this and the potential need for repeated applications, the procedure should be performed under general and regional anesthesia. The use of local anesthesia, as one of the anesthesia methods mentioned, is considered to be very low-risk and the least stressful overall.

Comparing the use of local anesthesia with the use of sedoanalgesia to perform the botulinum toxin A injection is equivalent to comparing two guideline-compliant standard treatments. The confirmation of our hypothesis, namely that performing the procedure under local anesthesia is equivalent to performing it under sedoanalgesia (non-inferiority study), could serve to optimize the treatment of overactive bladder patients and contribute to an increase in the level of health protection by strengthening the role of local anesthesia in the context of this procedure as an efficient option with the elimination of all anesthetic risks and as a first-choice procedure.

All patients with overactive bladder symptoms who fulfill the inclusion criteria and present at the Urogynecology Outpatient Clinic of the Department of Gynecology and Obstetrics at the LKH Hochsteiermark in Leoben within 24 months will be invited to participate in the study.

The following examinations are carried out on all patients before inclusion, in accordance with the examination standard of our department:

* Medical history: age, micturition frequency day/night, urinary leakage, sexuality, amount drunk, frequency of urinary tract infections, previous treatments for incontinence, parity, secondary diseases (diabetes mellitus, obesity, arterial hypertension, central nervous diseases, etc), previous gynecological operations, medication
* Urogynecological examination
* Urinalysis (midstream urine)
* Urodynamics with stress test
* Micturition protocol (will be scanned)
* Standardized questionnaires to assess incontinence symptoms and quality of life

This is an open prospective randomized controlled non-inferiority study. Patients participating in the study will be randomized into 2 arms (local anesthesia/sedoanalgesia) with a 1:1 ratio. Randomization will be done electronically (www.randomizer.at).

The sample design was calculated based on a non-inferiority study with pain score evaluation as the primary endpoint.

A sample size of 39 per group, including expected drop-outs (approximately 3 per group) results in a required number of participants of 84.

ELIGIBILITY:
Inclusion Criteria:

* Women with a minimum age of 18 years; no maximum age
* Unsuccessful conservative first and second-line treatment of OAB (defined as: completed pelvic floor/bladder training, local estrogenization of the vagina, at least one anticholinergic or ß3-mimetic oral therapy)
* Good German language skills

Exclusion Criteria:

* Pregnant women, breastfeeding women (no indication for approval)
* Women unable to give informed consent
* Refusal to participate in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — All individuals with anatomical organs of a woman
Enrollment: 84 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
pain assessed by numeric rating scale | twentyfour hours
  The numeric rating scale is a pain screening tool, commonly used to assess pain severity at that moment in time using a 0-10 scale, with zero meaning "no pain" and ten meaning "the worst pain imaginable".

SECONDARY OUTCOMES:
patient satisfaction assessed with postoperative anaesthesia questionnaire | twentyfour hours
  The postoperative anaesthesia questionnaire is a tool used to assess a patient's experience with anesthesia following surgery. It aims to gather information about the patient's perceptions of anesthesia-related outcomes and any adverse effects they may have experienced. It collects direct feedback from patients about their subjective experiences, including satisfaction and any discomfort or complications. Common sections and questions are about preoperative information, intraoperative experience, postoperative symptoms and overall satisfaction. Questions are answered with "yes" or "no".
quality of life assessed with King's Health Questionnaire | three and twelve months
  The King's Health Questionnaire is a disease specific, self-administered questionnaire designed to assess the impact of urinary incontinence on quality of life in women. The questions in this questionnaire are to be answered using a 0-4 scale, with zero meaning "not applicable" and four meaning "very accurate".

CONTACTS AND LOCATIONS:
Locations (1):
- LKH Hochsteiermark, Leoben, Austria

IPD SHARING:
Plan to Share IPD: No
The important and interesting data are published in a journal as part of the publication.

REFERENCES:
- [Background] Subramanian B, Shastri N, Aziz L, Gopinath R, Karlekar A, Mehta Y, Sharma A, Bapat JS, Jain P, Jayant A, Samra T, Perera A, Agarwal A, Shetty V, Bhatnagar S, Pandya ST, Jain P. ASSIST - Patient satisfaction survey in postoperative pain management from Indian subcontinent. J Anaesthesiol Clin Pharmacol. 2017 Jan-Mar;33(1):40-47. doi: 10.4103/joacp.JOACP_245_16. PMID 28413271
- [Background] Smith I, Avramov MN, White PF. A comparison of propofol and remifentanil during monitored anesthesia care. J Clin Anesth. 1997 Mar;9(2):148-54. doi: 10.1016/S0952-8180(96)00240-1. PMID 9075041
- [Background] Barba M, Lazar T, Cola A, Marino G, Manodoro S, Frigerio M. Learning Curve of Botulinum Toxin Bladder Injection for the Treatment of Refractory Overactive Bladder. Int J Womens Health. 2022 Jan 4;14:1-7. doi: 10.2147/IJWH.S345454. eCollection 2022. PMID 35018123
- [Background] Schurch B, Reitz A, Tenti G. Electromotive drug administration of lidocaine to anesthetize the bladder before botulinum-A toxin injections into the detrusor. Spinal Cord. 2004 Jun;42(6):338-41. doi: 10.1038/sj.sc.3101593. PMID 15007374
- [Background] Faure Walker N, Macpherson F, Tasleem A, Rampal T. Interventions to improve tolerability of local anesthetic intradetrusor Botulinum toxin injections: A systematic review. Neurourol Urodyn. 2023 Jan;42(1):23-32. doi: 10.1002/nau.25061. Epub 2022 Oct 23. PMID 36378811
- [Background] Cox L, Cameron AP. OnabotulinumtoxinA for the treatment of overactive bladder. Res Rep Urol. 2014 Jul 21;6:79-89. doi: 10.2147/RRU.S43125. eCollection 2014. PMID 25157339